CLINICAL TRIAL: NCT01590758
Title: A Randomized, Double-Blind, Multicenter, Superiority, Placebo-Controlled Phase 3 Study of Pexiganan Cream 0.8% Applied Twice Daily for 14 Days in the Treatment of Adults With Mild Infections of Diabetic Foot Ulcers
Brief Title: Pexiganan Versus Placebo Control for the Treatment of Mild Infections of Diabetic Foot Ulcers
Acronym: OneStep-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dipexium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DPX-305
Record Dates: First submitted 2012-04-27; First posted 2012-05-03 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-04

CONDITIONS: Diabetic Foot Infection
Keywords: Diabetic Foot Ulcer Infection
MeSH Terms: interventions — pexiganan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical placebo control (Placebo Comparator)
  Interventions: Drug: Topical placebo cream; Other: Standard wound care
- Topical pexiganan cream 0.8% (Experimental)
  Interventions: Drug: Topical pexiganan cream 0.8%; Other: Standard wound care

INTERVENTIONS:
Drug: Topical pexiganan cream 0.8% — 14 days of treatment
  Other Names: MSI-78
  Arms: Topical pexiganan cream 0.8%
Drug: Topical placebo cream — 14 days of treatment
  Arms: Topical placebo control
Other: Standard wound care — 14 days of treatment

SUMMARY:
The purpose of this study is to establish the clinical superiority and the safety of topical pexiganan cream 0.8% plus standard local wound care, as compared to placebo cream plus standard local wound care, in the treatment of mildly infected diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus.
2. Male or female at least 18 years old.
3. Subject must agree to adhere to all protocol procedures and return for all scheduled visits, and must be willing and able to provide written informed consent.
4. Subject is to be treated on an outpatient basis.
5. Full thickness ulcer or a partial thickness ulcer on the foot distal to the malleoli with a surface area ≥ 1 cm2 after the wound has undergone appropriate debridement.
6. Localized mild infection of the ulcer.
7. The diagnosis of mild infection must be confirmed immediately following debridement at Baseline.
8. Subject must have plain radiographs taken within 2 days prior to entry showing no evidence of bony abnormalities consistent with osteomyelitis, or gas compatible with tissue crepitus, in the affected foot.

Exclusion Criteria:

1. IDSA-defined moderate infection.
2. IDSA-defined severe infection.
3. Infected diabetic foot ulcer that is associated with local wound complications such as prosthetic materials or protruding surgical hardware.
4. > 1 infected foot ulcer.
5. Subject is currently receiving topical antimicrobial treatment for a localized infection of the study ulcer and whose infection is improving in response to treatment.
6. Subject has received a systemic antibiotic within 48 hours prior to Screening.
7. Concurrent or expected to require systemic antimicrobials during the study period for any infection, including diabetic foot ulcer.
8. Bone or joint involvement is suspected based on clinical examination or plain X-ray.
9. Clinically significant peripheral arterial disease requiring vascular intervention.
10. Subject is expected to be unable to care for the ulcer or return for all scheduled visits because of hospitalization, vacation, disability, etc. during the study period, or is unable to safely monitor the infection status at home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2014-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Silverman, MD, Study Director — BioStrategics Consulting Ltd
Locations (30):
- United States (30):
  - Birmingham, Alabama
  - Glendale, Arizona
  - Mesa, Arizona
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Bakersfield, California
  - Fair Oaks, California
  - Fresno, California
  - Los Angeles, California
  - Boynton Beach, Florida
  - Hialeah, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - South Miami, Florida
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Cambridge, Massachusetts
  - Missoula, Montana
  - Las Vegas, Nevada
  - Emerson, New Jersey
  - Greenville, North Carolina
  - Toledo, Ohio
  - Pittsburgh, Pennsylvania
  - Aiken, South Carolina
  - Baytown, Texas
  - Dallas, Texas
  - McAllen, Texas
  - McKinney, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited at outpatient clinics and practices
Pre-assignment Details: No wash-out or run-in periods; eligible subjects were immediately assigned to treatment
Groups:
- Topical Pexiganan Cream 0.8%: Topical pexiganan cream 0.8%: 14 days of treatment + 14 days of follow-up (28-day trial period)
  Standard wound care: 28-day trial period
- Topical Placebo Control: Topical placebo cream: 14 days of treatment + 14 days of follow-up (28-day trial period)
  Standard wound care: 28-day trial period
Period: Overall Study
Arm/Group | Topical Pexiganan Cream 0.8% | Topical Placebo Control
Started | 85 | 104
Completed | 80 | 97
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Topical Pexiganan Cream 0.8%: Topical pexiganan cream 0.8%: 14 days of treatment
  Standard wound care: 28-day trial period
- Topical Placebo Control: Topical placebo cream: 14 days of treatment
  Standard wound care: 28-day trial period
- Total: Total of all reporting groups
Arm/Group | Topical Pexiganan Cream 0.8% | Topical Placebo Control | Total
Number analyzed (Participants) | 85 | 104 | 189
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 59.22 (10.14) | 58.42 (10.97) | 58.78 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 31 | 53
  Male | 63 | 73 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 52 | 91
  Not Hispanic or Latino | 46 | 52 | 98
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 19 | 17 | 36
  White | 64 | 82 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 85 | 104 | 189
Wound surface area [Count of Participants; unit: Participants]
  <1 sq cm | 1 | 1 | 2
  1 - <2 sq cm | 41 | 52 | 93
  >=2 sq cm | 43 | 51 | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response
Description: The numbers of participants with Clinical Response, defined as resolution of infection, are reported.
Time Frame: 28 days
Population: Intent-To-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Pexiganan Cream 0.8% | Topical Placebo Control
Number analyzed (Participants) | 85 | 104
Participants | 43 | 63

2. Secondary Outcome: Number of Participants With Microbiological Success
Description: The numbers of participants with Microbiological Response, defined as eradication of all initial pathogens, are reported.
Time Frame: 28 days
Population: Intent-To-Treat Microbiological (positive for baseline pathogens)
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Pexiganan Cream 0.8% | Topical Placebo Control
Number analyzed (Participants) | 59 | 76
Participants | 16 | 28

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: The numbers of participants with TEAEs, including those with Serious TEAEs, are reported
Time Frame: 28 days
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Pexiganan Cream 0.8% | Topical Placebo Control
Number analyzed (Participants) | 85 | 104
Participants
  Incidence of any TEAE | 26 | 25
  Incidence of Serious TEAE | 9 | 3

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Topical Pexiganan Cream 0.8% | Topical Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/104
Serious Adverse Events (participants affected / at risk) | 9/85 | 3/104
Other Adverse Events (participants affected / at risk) | 6/85 | 4/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Pexiganan Cream 0.8% (N=85) | Topical Placebo Control (N=104)
Osteomyelitis (Infections and infestations) | 3 (3) | 0 (0)
Gangrene (Infections and infestations) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Diabetes inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Pexiganan Cream 0.8% (N=85) | Topical Placebo Control (N=104)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1)
Osteomyelitis (Infections and infestations) | 3 (3) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no multi-site publication within 18 months of study completion, Site shall have right to publish subject to: 1) Prior to submitting/presenting, Site shall provide Sponsor a copy; Sponsor shall have 60 days to review/comment. 2) Site shall remove any Confidential Information prior to submitting/presenting the materials. 3) Site shall further delay publication/presentation for up to 120 days to allow Sponsor to protect its interests in any Sponsor Inventions described in any such materials.